CLINICAL TRIAL: NCT00314197
Title: Study That Examines Integration of the Telephone Linked Care Behavioral Change (Automated Counseling) System Into Primary Care
Brief Title: Improving Health Behaviors Through Telephone Linked Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: American Academy of Family Physicians (Other)
Collaborators: Robert Wood Johnson Foundation (Other); Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 06-005
Record Dates: First submitted 2006-04-11; First posted 2006-04-13 (Estimated); Last update posted 2007-09-26 (Estimated); Status verified 2007-09

CONDITIONS: Diet; Physical Activity; Smoking; Alcohol Abuse
Keywords: automated counseling system; telephone-based intervention; behavior change
MeSH Terms: conditions — Motor Activity; Smoking; Alcoholism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Telephone Linked Care - Behavior Change Counseling System
Behavioral: Telephone-linked behavioral counseling

SUMMARY:
The investigators propose to conduct a randomized controlled trial at the patient level of the Telephone Linked Care - Behavioral Change (TLC-BC) system, which is designed to promote smoking cessation, reduce risky drinking, and improve physical activity and diet. They expect to:

1. successfully integrate an automated telephone behavior change intervention into primary care practices;
2. demonstrate improvement in health behaviors for individuals randomized (assigned by systematic chance) to use the TLC-BC system compared to individuals who receive written health education informational packets; and
3. evaluate the direct costs associated with the use and operation of the TLC-BC system.

Project aims and hypotheses follow:

Aim 1: Integrate a proven, totally automated computer telephone intervention, Telephone Linked Care - Behavior Change (TLC-BC), into primary care practices. This will be assessed by the patient and clinician/staff surveys at the end of data collection.

Aim 2: Demonstrate an improvement in health behaviors for individuals randomized to use the TLC-BC system compared to individuals who receive written informational packets.

Aim 3: Evaluate the direct costs associated with the use and operation of the TLC-BC system within the primary care setting.

Hypothesis 1: The Telephone Linked Care - Behavioral Change system will be successfully implemented by patients and practices.

Hypothesis 2: At 6 months a clinically significant improvement in behavioral change rates will be demonstrated for diet, physical activity, and smoking in the intervention group compared to patients in the control group.

Hypothesis 3: At baseline, 3, 6, and 9 months risky drinking will be identified, but there will be no difference in improvement between the study groups.

DETAILED DESCRIPTION:
See above

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Capable of giving informed consent
* Reliable access to a phone
* Able to read English

Exclusion Criteria:

* Less than 18 years of age
* Not capable of giving informed consent
* No reliable access to a phone
* Unable to read English (including blindness)
* Too ill to participate
* Not willing to allow the Telephone Linked Care - Behavior Change system to provide health information reports based on responses to physician

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2006-04; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
At 6 months a clinically significant improvement in behavioral change rates will be demonstrated for diet, physical activity and smoking in the intervention group compared to patients in the control group | 6 months
At baseline, 3, 6, and 9 months risky drinking will be identified, but there will be no difference in improvement between the study groups. | baseline, 3, 6, and 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Wilson D Pace, MD, FAAFP, Principal Investigator — American Academy of Family Physicians National Research Network
Locations (1):
- American Academy of Family Physicians National Research Network, Leawood, Kansas, United States